CLINICAL TRIAL: NCT04691414
Title: EXOMEDIANE - Retrospective Study Using High Throughput Sequencing (HTS) on Biological Samples to Improve Genetic Counseling for Patients With Previously Explored Craniofacial Midline Defects.
Brief Title: Retrospective Study Using Next Generation Sequencing (NGS) on Biological Samples to Improve Genetic Counseling for Patients With Previously Explored Craniofacial Midline Defects.
Acronym: EXOMEDIANE
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC20_8894_EXOMEDIANE
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Holoprosencephaly
MeSH Terms: conditions — Holoprosencephaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — national biobank
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: NGS — next-generation sequencing on preexisting samples

SUMMARY:
Holoprosencephaly, or HPE, is the most common congenital cerebral malformation in humans and the most severe of a group of pathologies related to a deficiency of the SHH signalling pathway (Sonic Hedgehog SHH-D). It is characterized by severe cerebral and craniofacial abnormalities.

The regulation of SHH concentration is therefore crucial for correct craniofacial development.

Despite the recent identification of about 20 genes, 70% of cases of EHPE and craniofacial midline abnormalities of genetic origin do not have a molecular diagnosis. It is therefore important to continue the search for new candidate genes to improve the understanding of brain and facial development and to improve genetic counseling for these families.

The development of Next-Generation Sequencing (NGS) technologies opens up the possibility of studying the exome or even the genome in a single manipulation. The latter type of analysis is particularly well suited to the discovery of new genes and will therefore improve the care of patients and their families.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Craniofacial Midline Facial Anomalies (CMFLA) collected for genetic analysis
* Patients and relatives for whom consent for research-related genetic testing is available. A "trio" - patient and both parents is required for analysis of variant segregation and determination of mode of transmission.
* For patients who are minors, parental authority(ies) who have given consent for research genetic testing.
* Affiliation to a social security scheme
* Patient and parents do not object to their participation in the research.
* In the case of a patient who has reached the age of majority since the initial consent was obtained, a patient who has given consent to proceed with genetic analyses for research purposes.

Exclusion Criteria:

* adults subject to legal protection (safeguard of justice, curatorship, guardianship), persons deprived of liberty.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 17 Trios : 17 patient with Craniofacial Midline Facial Anomalies and both parents already diagnosed in routine care. Blood samples for all trio must be available in the biobank and parents and patient if he's not a minor have to accept genetic analyses.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with an identified genetic abnormality | 6 months
  Number of patients with an identified genetic abnormality

SECONDARY OUTCOMES:
Number of new genes identified | 6 months
  Number of new genes identified, and possible recurrence of variants in one or more new genes of interest.
Pathogenic variants | 6 months
  Percentage of pathogenic variants identified in genes of the SHH pathway
Modes of transmission of pathogenic variants | 6 months
  Percentage of variants identified according to the different modes of transmission (de novo, autosomal dominant, X-linked, autosomal recessive, oligogenism)

CONTACTS AND LOCATIONS:
Overall Officials: Alinoë LAVILLAUREIX, Principal Investigator — CHU Rennes
Locations (1):
- CHU Rennes, Rennes, France

IPD SHARING:
Plan to Share IPD: No